CLINICAL TRIAL: NCT02703467
Title: Exhaled Hydrogen Sulphide as a Biomarker of Airways Disease in Asthma
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13/LO/1453
Record Dates: First submitted 2016-02-23; First posted 2016-03-09 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: Exhaled hydrogen sulphide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy subjects will have no significant medical history and no previous history of asthma or other serious illnesses. They should be non-smokers. The investigators willl measure spirometry and ensure that the values lie within the normal predicted range.
- Asthmatics: Patients diagnosed as having asthma will be recruited from Royal Brompton Hospital Asthma Clinics. These patients will have a range of severity of asthma ranging from mild-moderate to severe asthma patients. The diagnosis of asthma is ascertained as described in the inclusion criteria.

SUMMARY:
The purpose of this study will be to determine whether there is any role for measuring Hydrogen Sulphide (H2S) in the exhaled breath in terms of management of the patient with asthma.

The investigators will recruit patients with a range of severity of asthma and health volunteers. Levels of Hydrogen Sulphide will be measured in exhaled breath and blood. Also exhaled Nitric Oxide, Spirometry and asthma symptom scores will be measured at each study visit. Participants will attend either 2 or 4 separate visits.

The investigators will determine whether there is a relationship between exhaled Hydrogen Sulphide and asthma severity.

DETAILED DESCRIPTION:
Objectives:

1. Perform a cross-sectional study in non-asthmatic subjects and asthmatic subjects of varying severities of the levels of Hydrogen Sulphide in exhaled breath in relation to the severity and control of asthma
2. Compare the levels of exhaled Hydrogen Sulphide with exhaled Nitric Oxide.

We will recruit 30 health volunteers and 90 patients with a range of severity of asthma.

Particpants will attend for either 2 or 4 visits. At these visits the following measurements will be taken:

1. Exhaled Hydrogen Sulphide
2. Serum Hydrogen Sulphide

2. Exhaled Nitric Oxide 3. Spirometry 4. Asthma Symptom Score (ACQ)

The investigators will use a Hydrogen Sulphide UV fluorescent machine Model T101 (0-50 ppb to 0-20 ppm) (Cal-Bay Control Inc, USA) to measure directly on line exhaled breath Hydrogen Sulphide. This method has been used previously in normal people, but we will first determine whether there is an exhaled flow-dependence on the measurement of H2S levels. The investigators will use a hand-held Nitric Oxide machine (NO Breath) to measure Nitric Oxide in exhaled breath.

Subjects must have asthma according to one or more of the following criteria documented in the last 12 months:

1. Improvement in FEV1 (forced expiratory volume at one second) ≥ 12% and 200ml predicted after inhalation of 400 mcg salbutamol
2. Airway hyper-responsiveness (PC20 <8mg/ml)
3. Diurnal variation in PEF (peak expiratory flow): amplitude % mean of twice daily PEF > 8%
4. Decrease in pre-bronchodilator FEV1 >12% and >200mls within 4 weeks after tapering treatment with one or more of the following drugs: inhaled corticosteroids, oral corticosteroids, long-acting beta-agonists, long-acting beta-agonists and short-acting beta-agonists.

PLUS A history of wheeze occurring spontaneously or on exertion

ELIGIBILITY:
Inclusion Criteria:

All patients must be able to give informed consent. The definition of the severity of their asthma will be according to the GINA (Global Initiative for Asthma) guidelines dependent on the amount of therapy needed to control asthma. The investigators will also include at least 45 patients with severe asthma defined on the basis of: Uncontrolled asthma: three or more of the following features present in any week in the previous 4 weeks:

* Daytime symptoms more than twice per week
* Any limitation of activities
* Nocturnal symptoms once or more per week
* Need for reliever treatment more than twice per week
* Pre bronchodilator FEV1 <80% predicted or personal best OR
* Frequent severe exacerbations (≥2 per year) OR
* Require prescription of daily or alternate day oral corticosteroids (OCS) to achieve asthma control despite the prescription of high dose inhaled corticosteroids (>1000mcg fluticasone propionate daily or equivalent) or maintenance oral corticosteroids plus a long acting beta agonist or one other controller medication (for example anti-cholinergics, leukotriene receptor antagonists or theophylline).

Diagnosis of asthma for the asthma cohort: Subjects must have asthma according to one or more of the following criteria documented in the last 12 months

* improvement in FEV1 ≥ 12% and 200ml predicted after inhalation of 400 mcg salbutamol
* airway hyper-responsiveness (PC20 <8mg/ml)
* diurnal variation in PEF: amplitude % mean of twice daily PEF > 8%
* decrease in pre bronchodilator FEV1 >12% and >200mls within 4 weeks after tapering treatment with one or more of the following drugs: inhaled corticosteroids, oral corticosteroids, long-acting beta-agonists, long-acting beta-agonists and short-acting beta-agonists.

PLUS a history of wheeze occurring spontaneously or on exertion

Exclusion Criteria:

* Current smoker, or Ex-smoker with a >10 year pack history or having smoked within the past 6 months.
* Significant alternative diagnoses that may mimic or complicate asthma, in particular dysfunctional breathing, panic attacks, and overt psychosocial problems (if these are thought to be the major problem rather than in addition to severe asthma)
* Significant other primary pulmonary disorders in particular pulmonary embolism, pulmonary hypertension, interstitial lung disease and lung cancer
* Subjects with emphysema and bronchiectasis should only be excluded if this is thought to be the major pulmonary disorder rather than in addition to severe asthma
* Diagnosis or current investigation of occupational asthma
* Any subjects currently participating, or having participated within 3 months of the first dose in a study using a new molecular entity, or the first dose in any other study investigating drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit a cohort healthy subjects by advertisement within the Hospital and within the general public (by newspaper advertisement). The investigators will also recruit subjects with asthma from paients attending Asthma Clinics at the Royal Brompton and Harefiled NHS Trust.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian F Chung, MBBS MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy: Healthy participants
- Mild-moderate: Mild-moderate asthma patients
- Severe: Severe asthma patients
Period: Overall Study
Arm/Group | Healthy | Mild-moderate | Severe
Started | 20 | 5 | 45
Completed | 20 | 5 | 45
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy | Mild-moderate | Severe | Total
Number analyzed (Participants) | 20 | 5 | 45 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (3.5) | 55.6 (5.9) | 55.9 (11.5) | 54.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 3 | 31 | 47
  Male | 7 | 2 | 14 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 5 | 45 | 70

OUTCOME MEASURES:

1. Primary Outcome: Hydrogen Sulphide in Exhaled Breath
Description: Level of hydrogen sulphide in exhaled breath measured as parts per billion
Time Frame: At baseline visit
Measure: Mean (Standard Error); unit: parts per billion
Arm/Group | Healthy | Mild-moderate | Severe
Number analyzed (Participants) | 20 | 5 | 45
parts per billion | 5.0 (0.6) | 3.2 (1.0) | 4.9 (1.3)
Statistical Analysis 1: Comparison: Healthy vs Severe; Test type: Superiority; p > 0.05, t-test, 2 sided — calculated

2. Secondary Outcome: FEV1
Description: Forced expiratory volume in one second as percent of predicted value (%)
Time Frame: At baseline visit
Measure: Mean (Standard Error); unit: per cent of predicted value
Groups:
- Healthy Subjects: Healthy participants
- Mild-moderate Asthma: Participants with Mild-moderate asthma
- Severe Asthma: Participant with Severe asthma
Arm/Group | Healthy Subjects | Mild-moderate Asthma | Severe Asthma
Number analyzed (Participants) | 20 | 5 | 45
per cent of predicted value | 98.9 (4.1) | 92.0 (11.1) | 73.6 (4.3)

3. Secondary Outcome: FVC (Forced Vital Capacity)
Description: Forced vital capacity as per cent of predicted
Time Frame: At 4 visits which occur during the study duration, up to 1 year
Measure: Mean (Standard Error); unit: per cent of predicted value (%)
Arm/Group | Healthy | Mild-moderate | Severe
Number analyzed (Participants) | 20 | 5 | 45
per cent of predicted value (%) | 105.1 (4.3) | 97.40 (15.3) | 88.22 (3.5)

4. Secondary Outcome: Exhaled Nitric Oxide
Description: Levels of nitric oxide in exhaled breath in parts per billion
Time Frame: At 4 visits which occur during the study duration, up to 1 year
Measure: Mean (Standard Error); unit: parts per billion
Groups:
- Severe Asthma: Participants with severe asthma
Arm/Group | Healthy Subjects | Mild-moderate Asthma | Severe Asthma
Number analyzed (Participants) | 20 | 5 | 45
parts per billion | 25.41 (6.3) | 39.42 (13.6) | 39.45 (2.2)

5. Secondary Outcome: Blood Hydrogen Sulpide Level
Description: Hydrogen Sulpide level measurements from blood
Time Frame: At 4 visits which occur during the study duration, up to 1 year
Population: Data not collected
Arm/Group | Healthy Subjects | Mild-moderate Asthma | Severe Asthma
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Healthy | Mild-moderate | Severe
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/5 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/5 | 0/45
Other Adverse Events (participants affected / at risk) | 0/20 | 0/5 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes